CLINICAL TRIAL: NCT06043050
Title: Sequential Predictions Under Repeated Interventions: Estimating the Risk of Major Bleeding or Death With and Without Prophylactic Platelet Transfusion in Thrombocytopenic Neonates.
Brief Title: PRedicting OutcomeS in Preterm nEonates With thromboCyTopenia
Acronym: PROSPECT
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Sanquin Research & Blood Bank Divisions (Other); Amsterdam University Medical Center (Other)
Responsible Party: Principal Investigator, Hilde van der Staaij, MD, MD, Coordinating Investigator, Leiden University Medical Center
Other Study IDs: 22-3028
Record Dates: First submitted 2023-08-17; First posted 2023-09-21 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Thrombocytopenia; Intraventricular Hemorrhage; Platelet Transfusion
Keywords: Sequential prediction under interventions; Causal prediction; Hemorrhage; Neonate; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune; Hemorrhage; Thrombocytopenia | interventions — Platelet Count; Platelet Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neonates with severe thrombocytopenia: Neonates with a gestational age below 34 weeks and at least one platelet count below 50x10^9/L, who were admitted to a NICU between January 1st, 2017 and January 1st, 2022.
  Interventions: Drug: Platelets

INTERVENTIONS:
Drug: Platelets — Observational data: all platelet transfusions recorded in routine care medical file data.
  Other Names: Platelet transfusion

SUMMARY:
Preterm neonates often receive platelet transfusions when their platelet count is low to prevent bleeding. However, it is currently unclear which infants benefit from such transfusions. A recent randomized controlled trial (PlaNeT-2/MATISSE trial) showed that the higher platelet count threshold for transfusion was associated with a higher risk of major bleeding or death. Current transfusion protocols are based only on platelet count thresholds. However, neonates with similar platelet counts may have different bleeding risks due to varying clinical conditions. There is an important unmet medical need to identify which neonates with low platelet counts (i.e., severe thrombocytopenia) will benefit from a transfusion. Ideally, clinicians would be able to repeatedly predict a neonate's risk of major bleeding or death with and without giving a platelet transfusion, taking into account the neonate's clinical condition at that particular time. Obtaining personalized risk estimates under specific treatment strategies, with updated predictions at each new treatment decision moment, is called 'sequential prediction under interventions'. The investigators set up an international multicenter observational cohort study to develop a model to predict major bleeding or death with and without platelet transfusion at any time point during the first week after the onset of severe thrombocytopenia. This model is designed to support platelet transfusion decisions in the NICU and may help clinicians balance the benefits and harms of platelet transfusion based on updated characteristics of the neonate at the time of prediction.

DETAILED DESCRIPTION:
Main objective: To develop a sequential interventional prediction model to support transfusion decisions by predicting the risk of major bleeding or death with and without giving a platelet transfusion to neonates with severe thrombocytopenia (i.e., platelet count below 50x10^9/L), conditional on their characteristics present at the moment of prediction.

Study design: Multicenter international observational cohort study.

Study population: Neonates with a gestational age below 34 weeks and at least one platelet count below 50x10^9/L, admitted to a neonatal intensive care unit (NICU) between January 1st 2017 and January 1st 2022.

Main study endpoint: Major bleeding or mortality during NICU admission

Assessments: Only routine care data will be collected. This includes platelet counts and transfusions, cranial (head) ultrasounds and other information on bleeding, and multiple clinical variables.

Statistical analyses: Development of a sequential prediction model under interventions using the cloning-censoring-weighting approach with inverse probability weighting. Validation of the model in a separate cohort of preterm neonates with severe thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age at birth <34 weeks;
2. At least one platelet count <50x109/L;
3. Admission to a participating tertiary care NICU, including postnatal transfers, between January 1st, 2017 and January 1st, 2022.

Exclusion Criteria:

1. A severe congenital malformation;
2. Only spurious platelet counts <50x109/L (e.g. clots in the sample, or a very rapid recovery to a normal platelet count without platelet transfusion);
3. Only platelet counts <50x109/L in the context of exchange transfusion;
4. Major intracranial bleeding prior to the onset of severe thrombocytopenia. Neonates with major bleeding after the end of follow-up will not be excluded, but will be recorded as having had no major bleeding during the study.

Ages: 22 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with a gestational age below 34 weeks and at least one platelet count below 50x10^9/L, admitted to a NICU between January 1st, 2017 and January 1st, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 1042 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
A composite of major bleeding or death during NICU admission is the primary outcome. Neonates who first had a major bleeding and then died reach the endpoint at the time of the major bleeding. | From onset of severe thrombocytopenia until one week thereafter. The risk of major bleeding or death is predicted within 3 days and within 14 days from each moment of prediction during this time frame.
  The investigators defined major bleeding as either one of the following:
  1. Intraventricular hemorrhage (IVH) grade 3 or IVH of any grade in combination with parenchymal involvement (according to the Volpe grading system);
  2. Parenchymal hemorrhage (without IVH) or cerebellar hemorrhage (>4 mm visible on cranial ultrasound, not if ≤4 mm visible on MRI only);
  3. Pulmonary hemorrhage, defined as a fresh bleed from the trachea requiring intubation or ventilation, or a fresh bleed from the tube requiring increased ventilatory requirements;
  4. Any type of severe hemorrhage, including gastrointestinal bleeding, if associated with hemodynamic instability (e.g., hypotension) and/or requiring one of the following interventions within 24h*:
     1. Red blood cell transfusion
     2. Volume boluses
     3. Inotropes (either start of inotropes, or increased dose of current therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Hilde van der Staaij, MD, Study Director — Leiden University Medical Center and Sanquin Blood Supply Foundation; Johanna G van der Bom, MD/PhD/Prof, Principal Investigator — Leiden University Medical Center; Camila Caram-Deelder, MSc/PhD, Principal Investigator — Leiden University Medical Center; Enrico Lopriore, MD/PhD/Prof, Principal Investigator — Leiden University Medical Center; Karin Fijnvandraat, MD/PhD/Prof, Principal Investigator — Amsterdam University Medical Center; Suzanne F Fustolo-Gunnink, MD/PhD, Principal Investigator — Sanquin Blood Supply Foundation; Wes Onland, MD/PhD, Principal Investigator — Amsterdam University Medical Center; Nan van Geloven, MSc/PhD, Principal Investigator — Leiden University Medical Center; Ilaria Prosepe, MSc, Principal Investigator — Leiden University Medical Center
Locations (12):
- Charité - Universitätsmedizin Berlin, Berlin, Metropolregion Berlin-Brandenburg, Germany
- Netherlands (10):
  - Radboud University Medical Center, Amalia Children's hospital, Nijmegen, Gelderland
  - Maastricht University Medical Center, MosaKids, Maastricht, Limburg
  - Máxima Medical Center, Veldhoven, North Brabant
  - Amsterdam University Medical Center, Emma Children's hospital, location VUmc, Amsterdam, North Holland
  - Amsterdam University Medical Center, Emma Children's hospital, location AMC, Amsterdam, North Holland
  - Isala clinics, Zwolle, Overijssel
  - University Medical Center Groningen, Beatrix Children's hospital, Groningen, Provincie Groningen
  - Leiden University Medical Center, Willem Alexander Children's hospital, Leiden, South Holland
  - Erasmus University Medical Center, Sophia pediatric hospital, Rotterdam, South Holland
  - University Medical Center Utrecht, Wilhelmina Children's hospital, Utrecht, Utrecht
- Karolinska University Hospital, Stockholm, Södermanland and Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to the sensitivity of the data, the underlying data sets will not be shared publicly due to ethical/privacy restrictions. However, all analyses will be documented, reproducible and available for audit. The data dictionary will be available upon request or as appendix in the manuscript. We might consider restricted access to the raw data in a repository when the target journal deems this necessary for publication. For future collaboration with the research partners or for data transfer/sharing, written agreements on data management, privacy, data ownership and intellectual properties will be made, such as a research collaboration agreement and data sharing agreement, and discussed with the support of Legal/Privacy/RDM experts where appropriate. In line with the Netherlands Code of Conduct for Research Integrity, raw and processed will be stored for a period of at least 10 years. The LUMC has long-term storage with back-up available for this.

REFERENCES:
- [Background] Curley A, Stanworth SJ, Willoughby K, Fustolo-Gunnink SF, Venkatesh V, Hudson C, Deary A, Hodge R, Hopkins V, Lopez Santamaria B, Mora A, Llewelyn C, D'Amore A, Khan R, Onland W, Lopriore E, Fijnvandraat K, New H, Clarke P, Watts T; PlaNeT2 MATISSE Collaborators. Randomized Trial of Platelet-Transfusion Thresholds in Neonates. N Engl J Med. 2019 Jan 17;380(3):242-251. doi: 10.1056/NEJMoa1807320. Epub 2018 Nov 2. PMID 30387697
- [Background] Davenport P, Sola-Visner M. Hemostatic Challenges in Neonates. Front Pediatr. 2021 Mar 2;9:627715. doi: 10.3389/fped.2021.627715. eCollection 2021. PMID 33738269
- [Background] Davenport PE, Wood TR, Heagerty PJ, Sola-Visner MC, Juul SE, Patel RM. Platelet Transfusion and Death or Neurodevelopmental Impairment in Children Born Extremely Preterm. JAMA Netw Open. 2024 Jan 2;7(1):e2352394. doi: 10.1001/jamanetworkopen.2023.52394. PMID 38261320
- [Background] Fustolo-Gunnink SF, Fijnvandraat K, van Klaveren D, Stanworth SJ, Curley A, Onland W, Steyerberg EW, de Kort E, d'Haens EJ, Hulzebos CV, Huisman EJ, de Boode WP, Lopriore E, van der Bom JG; PlaNeT2 and MATISSE collaborators. Preterm neonates benefit from low prophylactic platelet transfusion threshold despite varying risk of bleeding or death. Blood. 2019 Dec 26;134(26):2354-2360. doi: 10.1182/blood.2019000899. PMID 31697817
- [Background] Fustolo-Gunnink SF, Fijnvandraat K, Putter H, Ree IM, Caram-Deelder C, Andriessen P, d'Haens EJ, Hulzebos CV, Onland W, Kroon AA, Vijlbrief DC, Lopriore E, van der Bom JG. Dynamic prediction of bleeding risk in thrombocytopenic preterm neonates. Haematologica. 2019 Nov;104(11):2300-2306. doi: 10.3324/haematol.2018.208595. Epub 2019 Feb 28. PMID 30819913
- [Background] Hernan MA, Wang W, Leaf DE. Target Trial Emulation: A Framework for Causal Inference From Observational Data. JAMA. 2022 Dec 27;328(24):2446-2447. doi: 10.1001/jama.2022.21383. PMID 36508210
- [Background] Keogh RH, Van Geloven N. Prediction Under Interventions: Evaluation of Counterfactual Performance Using Longitudinal Observational Data. Epidemiology. 2024 May 1;35(3):329-339. doi: 10.1097/EDE.0000000000001713. Epub 2024 Apr 18. PMID 38630508
- [Background] van der Staaij H, Stanworth SJ, Fustolo-Gunnink SF. Prophylactic Platelet Transfusions: Why Less Is More. Clin Perinatol. 2023 Dec;50(4):775-792. doi: 10.1016/j.clp.2023.07.007. Epub 2023 Aug 31. PMID 37866847
- [Background] van Geloven N, Swanson SA, Ramspek CL, Luijken K, van Diepen M, Morris TP, Groenwold RHH, van Houwelingen HC, Putter H, le Cessie S. Prediction meets causal inference: the role of treatment in clinical prediction models. Eur J Epidemiol. 2020 Jul;35(7):619-630. doi: 10.1007/s10654-020-00636-1. Epub 2020 May 22. PMID 32445007